CLINICAL TRIAL: NCT02091180
Title: Effect of Preoperative Mannitol Infusion on Cerebral Oxygen Saturation and Patients' Recovery After Laparoscopic Cholecystectomy
Brief Title: Mannitol Improves Cerebral Oxygen Saturation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Hany A. Mowafi, Associate professor, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012069
Record Dates: First submitted 2014-03-15; First posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Anesthesia
Keywords: Anesthesia; Recovery; laparoscopy; cholecystectomy
MeSH Terms: interventions — Mannitol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mannitol (Experimental): Patients will receive 0.5g/kg of 20% intravenous (i.v.) mannitol infusion over 10 minutes immediately before induction of anesthesia
  Interventions: Drug: Mannitol
- Control (Placebo Comparator): Patients will receive normal saline
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Mannitol — 0.5g/kg of 20% intravenous (i.v.) mannitol infusion over 10 minutes immediately before induction of anesthesia
  Other Names: mannite or manna sugar
  Arms: Mannitol
Drug: Control — Saline infusion
  Other Names: Saline
  Arms: Control

SUMMARY:
Decreased cerebral oxygen saturation (rSO2) was reported to occur during insufflation for laparoscopic procedures due to increased Intracranial pressure (ICP) with resultant decrease in cerebral perfusion pressure.

DETAILED DESCRIPTION:
Forty patients scheduled for laparoscopic cholecystectomy will be enrolled in this double blind, randomized controlled study. Patients will receive either 0.5g/kg of 20% intravenous (i.v.) mannitol infusion over 10 minutes immediately before induction of anesthesia (group M) or an equal volume of 0.9% normal saline instead (group C). Primary outcome measure is rSO2. Secondary outcome variables include extubation time, clinical assessment of consciousness recovery using the modified Observer's assessment of alertness/sedation scale (OAA/S) and the mini-mental state examination (MMSE) for cognitive evaluation after recovery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II
* aged between 25 and 50 years
* with a body mass index (BMI) 22-34 kg/m2

Exclusion Criteria:

* obstructive or restrictive pulmonary disease
* cardiac dysfunction

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
rSO2 | participants will be followed for the duration of surgery, an expected average of 1 hour

SECONDARY OUTCOMES:
extubation time | intraoperative
  time from end of anesthesia to fulfilling extubation criteria

OTHER OUTCOMES:
OAA/S | after surgery 30 minutes.
  alertness/sedation scale

CONTACTS AND LOCATIONS:
Overall Officials: Hany A Mowafi, MD, Study Director — Imam Abdulrahman Bin Faisal University
Locations (2):
- Saudi Arabia (2):
  - Anesthesia Department, University of Dammam, Khobar, EP
  - King Fahd Hosital of the University, Khobar, EP